CLINICAL TRIAL: NCT00415259
Title: Effects of Shoes Insoles on Symptoms and Disease Progression in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Principal Investigator, Kim Bennell, Professor Kim Bennell, University of Melbourne
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 350297
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laterally wedged shoe insoles (Experimental): Full-length 5 degree lateral wedged insoles worn inside the shoes daily for 12 months
  Interventions: Device: Laterally wedged shoe insoles
- Flat control insoles (Other)
  Interventions: Device: Control insole group

INTERVENTIONS:
Device: Laterally wedged shoe insoles — Full-length 5 degree lateral wedged insoles worn inside the shoes daily for 12 months
  Arms: Laterally wedged shoe insoles
Device: Control insole group — Flat control insoles worn inside the shoes daily for 12 months
  Arms: Flat control insoles

SUMMARY:
It is hypothesised that laterally wedged insoles will result in reduced knee pain and cartilage volume loss after 12 months of wear, compared to control insoles. People with symptomatic knee osteoarthritis will be recruited from the community and randomised to wear either laterally wedged insoles or control insoles for 12 months. Patients will be assessed at baseline and at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility will be confirmed by radiographic and clinical examination
* People with medial tibiofemoral joint OA fulfilling American College of Rheumatology classification criteria and reporting average knee pain on walking >3 on an 11-point scale
* varus knee malalignment on standing anteroposterior lower limb x-ray.

Exclusion Criteria:

* advanced radiographic knee OA (Kellgren and Lawrence stage 4
* knee surgery or intra-articular corticosteroid injection within 6 months
* current or past (within 4 weeks) oral corticosteroid use
* systemic arthritic conditions
* history of tibiofemoral/patellofemoral joint replacement or tibial osteotomy
* any other muscular, joint or neurological condition affecting lower limb function
* ankle/foot pathology or pain that precludes the use of insoles
* use of foot orthotics within past 6 months and
* use of footwear that does not accomodate an insole.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2005-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Knee pain via a visual analogue scale | Measured at baseline and 12 months
Disease progression via MRI measurements of knee cartilage volume | Measured at baseline and 12 months

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities (WOMAC) Oestoarthritis Index | Measured at baseline and 12 months
Patient perceived response to treatment | Measured at baseline and 12 months.
Health-related quality-of-life (via SF-36, AQoL questionnaires) | Measured at baseline and 12 months
Recorded use of health care | Measured at baseline and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kim Bennell, PhD, Principal Investigator — University of Melbourne
Locations (1):
- Centre for Health Exercise & Sports Medicine, School of Physiotherapy, The University of Melbourne, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Bennell KL, Bowles KA, Payne C, Cicuttini F, Williamson E, Forbes A, Hanna F, Davies-Tuck M, Harris A, Hinman RS. Lateral wedge insoles for medial knee osteoarthritis: 12 month randomised controlled trial. BMJ. 2011 May 18;342:d2912. doi: 10.1136/bmj.d2912. PMID 21593096
- [Derived] Bennell K, Bowles KA, Payne C, Cicuttini F, Osborne R, Harris A, Hinman R. Effects of laterally wedged insoles on symptoms and disease progression in medial knee osteoarthritis: a protocol for a randomised, double-blind, placebo controlled trial. BMC Musculoskelet Disord. 2007 Sep 24;8:96. doi: 10.1186/1471-2474-8-96. PMID 17892539